CLINICAL TRIAL: NCT05549128
Title: Effect of Transcutaneous Photobiomodulation on the Control of Chilhood Anxiety in Dental Care: Double- Blind Randomized Clinical Trial.
Brief Title: Transcutaneous Photobiomodulation on the Control of Chilhood Anxiety in Dental Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPMBAnx
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Anxiety
Keywords: anxiety; photobiomodulation
MeSH Terms: conditions — Anxiety Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: 2 groups: experimental group (G1), control group or placebo (G2) where ILIB and placebo will be applied respectively.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be performed for the application of the ILIB during the clinical session. An operator will be trained who will be the one who will perform the application. Another operator, in this case the researcher (blind), will be in charge of collecting the parameters to be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photobiomodulation (Experimental): laser therapy application for 10 minutes
  Interventions: Device: Photobiomodulation
- Sham photobiomodulation (Sham Comparator): sham laser therapy application for 10 minutes
  Interventions: Device: Photobiomodulation sham

INTERVENTIONS:
Device: Photobiomodulation — The red laser (DMC) will be applied with the aim of reducing the anxiety of children during the dental consultation. It will be continuously and directly with 60J of energy, wavelength of 660nm and 100mW/cm2 of power. The application will be located in the unilateral radial artery for 10 minutes. The laser will be transmitted through an appropriate bracelet where the laser tip fits perfectly. It is a painless, non-invasive method that does not cause any discomfort during application.
  Arms: photobiomodulation
Device: Photobiomodulation sham — The red laser (DMC) will be applied off. I
  Arms: Sham photobiomodulation

SUMMARY:
The objective of this study is to investigate whether photobiomodulation helps, collaborates, in the management of the child's anxiety in the dental office.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is a chronic psychiatric condition characterized by a widespread and disproportionate concern for adverse life circumstances and the anticipated occurrence of catastrophic and dramatic events. Often, the challenges of everyday life, whether potential or real, are feared, as they are expected to increase and lead to irreparable consequences. Currently photobiomodulation is a practice used in many areas of health successfully. In the area of anxiety disorders has shown very promising results improving patient behavior. If we understand that photobiomodulation is a non-invasive therapy and with enough evidence of its safety, we must investigate to complement traditional behavioral management techniques. The objective of this study is to investigate whether photobiomodulation (ILIB) helps, collaborates, in the management of the child's anxiety in the dental office.

The sample will be selected from the assistance centers that have an agreement with UCU, Federico Ozanam School, San José College, UCU University Health Clinic. Participants will be randomly distributed into 2 groups: experimental group (G1), control group or placebo (G2) where ILIB and placebo will be applied respectively. It will be evaluated in level of anxiety by: Facial Image Scale (FIS) and the Venham Imaging Test (VPT) in the conditioned room prior to dental care (16)(17). Physiological parameters will also be measured: blood pressure, oximetry, heart rate, pulse, weight, height. ILIB applications will be carried out in 2 clinical sessions with an interval between them of at least 48hrs.

ELIGIBILITY:
Inclusion Criteria:

Children 6 and 12 years old. Children who do not consume oral anxiolytics. Children who need dental treatment. Children whose responsible adults have accepted informed consent. Children who have signed a nod of care.

Exclusion Criteria:

Children who are taking medications that alter the central nervous system ( Children with psychiatric or psychological disorders. Children with motor disorders such as cerebral palsy. Patients who do not fall into the age range of inclusion. Patients whose responsible adults do not agree to sign the informed consent. Children who do not give their assent to attention.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 30 minutes
  Facial Image Scale (FIS) in the conditioned room prior to dental care.

SECONDARY OUTCOMES:
heart rate | 30 minutes
  The oximeter will be used in this work to measure the heart rate of children before and after dental treatment. The device will be placed on a finger of the child's hand, it is note worthy that it is a device or that it does not cause any type of discomfort.

IPD SHARING:
Plan to Share IPD: No